CLINICAL TRIAL: NCT00985660
Title: Single-Dose Fasting Bioequivalence Study of Nisoldipine Extended-Release Tablets (30 mg; Mylan) and Sular® Extended Release Tablets (30 mg; First Horizon) in Healthy Volunteers
Brief Title: Bioequivalence Study of Nisoldipine Extended-Release Tablets, 30 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Wayne Talton, Vice President, Regulatory Affairs, Mylan Pharmaceuticals Inc.
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NISO-0752
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Healthy

ARMS (2):
- Test: (Experimental): Nisoldipine ER Tablets, 30 mg
  Interventions: Drug: Nisoldipine Extended-release Tablets, 30 mg
- Reference (Active Comparator): Sular Extended-release Tablets, 30 mg
  Interventions: Drug: Sular® Extended Release Tablets, 30 mg

INTERVENTIONS:
Drug: Nisoldipine Extended-release Tablets, 30 mg — 1 x 30 mg Tablet under fasting conditions
  Arms: Test:
Drug: Sular® Extended Release Tablets, 30 mg — 1 x 30 mg Tablet under fasting conditions
  Arms: Reference

SUMMARY:
The objective of this study was to investigate the bioequivalence of nisoldipine extended-release 30 mg tablets (by Mylan Pharmaceuticals Inc.) with Sular® Extended-Release 30 mg tablet (manufactured for First Horizon) following a single, oral 30 mg (1 × 30 mg tablet) dose administration in healthy adult subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older.
* Sex: Male and/or non-pregnant, non-lactating female.

  * Women of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 21 days prior to the start of the study and on the evening prior to each dose administration. If dosing is scheduled on Sunday or Monday, the HCG pregnancy test should be given within 48 hours prior to dosing for each study period. An additional serum (β-HCG) pregnancy test will be performed upon completion of the study.
  * Women of childbearing potential must practice abstinence or be using an acceptable form of contraception throughout the duration of the study. No hormonal contraceptives or hormonal replacement therapies are permitted in this study. Acceptable forms of contraception include the following:

    1. Intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
    2. Barrier methods containing or used in conjunction with a spermicidal agent, or
    3. Surgical sterilization
  * Women will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

    1. Postmenopausal with an absence of menses for at least one (1) year, or
    2. Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
    3. Total hysterectomy
  * During the course of the study, from study screen until study exit - including the washout period, all men and women of childbearing potential must use a spermicide containing barrier method of contraception in addition to their current contraceptive method. This advice should be documented in the informed consent form.
* Weight: At least 60 kg (132 lbs) for men and 48 kg (106 lbs) for women with all subjects having a Body Mass Index (BMI) less than or equal to 30 but greater than or equal to 19.
* All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, Hepatitis B and Hepatitis C tests, HIV test, 12-lead ECG, and urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiates, phencyclidine, and methadone) performed within 21 days of the initial dose of study medication

Exclusion Criteria:

* Institutionalized subjects will not be used.
* Social Habits:

  * Use of any tobacco-containing products within 1 year of the start of the study.
  * Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
  * Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
  * Any recent, significant change in dietary or exercise habits.
  * A positive test for any drug included in the urine drug screen.
  * History of drug and/or alcohol abuse.
* Medications:

  * Use of any prescription or over-the-counter (OTC) medications within the 14 days prior to the initial dose of study medication.
  * Use of any hormonal contraceptives or hormone replacement therapy within 3 months prior to study medication dosing.
  * Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
* Diseases:

  * History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, or neurologic disease.
  * Acute illness at the time of either the pre-study medical evaluation or dosing.
  * A positive HIV, hepatitis B, or hepatitis C test.
* Abnormal and clinically significant laboratory test results:

  * Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
  * Abnormal and clinically relevant ECG tracing.
* Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
* Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
* Allergy or hypersensitivity to nisoldipine, any of the inactive ingredients, or other calcium channel blocker products.
* History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
* Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.
* Average sitting pulse rate less than 55 beats per minute after a five minute rest at screening OR prior to Period I Day 1 dosing. Pulse rate measurements will be taken in triplicate with at least two (2) minutes elapsing in-between measurements.
* Average sitting systolic blood pressure less than 90 mmHg or average sitting diastolic blood pressure less than 60 mmHg following a five (5) minute rest at screening OR prior to Period I Day 1 dosing. Blood pressure measurements will be taken in triplicate with at least two (2) minutes elapsing in-between readings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve | Serial plasma samples collected for up to 72 hours post-dose
Maximum Plasma Concentration | Serial plasma samples collected up to 72 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc - Clinical Trial Results — http://www.mpibiostudies.com